CLINICAL TRIAL: NCT00695188
Title: Methotrexate Polyglutamate Levels as a Marker for the Clinical Outcome in the Treatment of Rheumatoid Arthritis A Multicenter, Randomized, Double-blind, Controlled Phase IV Trial
Brief Title: Methotrexate Polyglutamate Levels as a Marker for the Clinical Outcome in the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ludwig-Boltzmann Institut fuer Rheumatologie, Balneologie und Rehabilitation (Other)
Responsible Party: Prim. Univ.-Prof. Dr. Hans Broell, Ludwig-Boltzmann Institut fuer Rheumatologie und Balneologie
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROMTX2007_01; EudraCT: 2007-006288-56
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Results first posted 2011-02-15 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2009-08

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; MTX polyglutamates; clinical outcome
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard dose (Other): Escalating dose
  Interventions: Drug: methotrexate
- High dose (Active Comparator): 25 mg
  Interventions: Drug: methotrexate

INTERVENTIONS:
Drug: methotrexate — oral administration Escalating dose (15, 20, 25 mg)
  Arms: Standard dose
Drug: methotrexate — 25 mg oral administration
  Arms: High dose

SUMMARY:
The primary objective is to determine whether erythrocyte polyglutamate levels are associated with objective clinical response in patients with rheumatoid arthritis after oral administration of low-dose methotrexate.The secondary aim of this study is to compare the efficacy and safety of standard dose methotrexate versus a higher starting dose.

DETAILED DESCRIPTION:
The folate antagonist methotrexate (MTX) is currently one of the most widely used drugs for the treatment of rheumatoid arthritis (RA).Although MTX is very effective and well tolerated, the major drawback is the large interpatient variability in the clinical response.MTX is intracellularly converted by folylpolyglutamate synthetase (FPGS) to methotrexate polyglutamates (MTXPGs), which enhance the intracellular retention of MTX. Furthermore, the γ-linked sequential addition of glutamic acid residues inhibits finals steps in the de novo purine and pyrimidine biosynthesis, resulting in anti-proliferative and anti-inflammatory effects.76 adult, MTX-naive patients who fulfill the American College of Rheumatology criteria (ACR) for RA with a Disease Activity Score in 28 joints (DAS-28) > 3.2 are enrolled at two sites in Vienna (Austria).Clinical status is assessed by the number of joint counts and the Health Assessment Questionnaire (HAQ).Patients are randomly assigned to receive either a standard dose or a higher starting dose of 25 mg orally. In week 5, a subcutaneous dose of 25 mg is administered to each patient to get a reference level (bioavailability of 100%).The patients participate for 16 weeks, in which blood samples are collected at weeks 1, 2, 5, 6, 10 and 11 to perform pharmacokinetic analyses and metabolite measurements.The determination of erythrocyte MTXPG-levels is performed by using a HPLC technique.The primary outcome is the objective clinical response (measured in a rheumatic score, DAS-28), secondary outcome parameters are quality of life and routine laboratory parameters used in rheumatology. This clinical outcome will be correlated with MTX pharmacokinetics in blood, MTXPG kinetics in erythrocytes, and their impact on the folate pathway.

ELIGIBILITY:
Inclusion Criteria:

* MTX-naive
* Age > 18 years
* DAS-28 > 3.2
* American College of Rheumatology-criteria for RA
* Chest-X-ray
* Informed consent
* Prednisolon < 10 mg a day

Exclusion Criteria:

* Pregnancy
* Lactation
* Renal and hepatic impairment
* Malignant diseases (last 5 years)
* Contraindications
* Human Immunodeficiency Virus (HIV), Hepatitis B and C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Broell, Prof. Dr., Principal Investigator — Ludwig-Boltzmann-Institut fuer Rheumatologie und Balneologie
Locations (2):
- Austria (2):
  - Kaiser-Franz-Josef-Spital, Vienna
  - Rheumazentrum Wien Oberlaa, Vienna

REFERENCES:
- [Derived] Hobl EL, Mader RM, Jilma B, Duhm B, Mustak M, Broll H, Hogger P, Erlacher L. A randomized, double-blind, parallel, single-site pilot trial to compare two different starting doses of methotrexate in methotrexate-naive adult patients with rheumatoid arthritis. Clin Ther. 2012 May;34(5):1195-203. doi: 10.1016/j.clinthera.2012.03.059. Epub 2012 Apr 18. PMID 22516039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were included at the outpatient unit of the Kaiser-Franz-Josef-Hospital, Department for Rheumatology, if they fulfilled the inclusion criteria
Groups:
- Standard Dose: Escalating dose (Start with 15 mg MTX/week, escalating dose until 25 mg/week, administered orally)
- High Dose: Start with 25 mg MTX per week, administered orally
Period: Overall Study
Arm/Group | Standard Dose | High Dose
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose | High Dose | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 6 | 4 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (15) | 62 (7) | 56 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Austria | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: DAS-28 (Disease Activity Score in 28 Joints)
Description: DAS stands for "Disease Activity Score" and is a measure of the activity of rheumatoid arthritis. In Europe the DAS is the recognized standard in research and clinical practice.
  The following parameters are included in the calculation:
  * Number of joints tender to the touch (TEN)
  * Number of swollen joints (SW)
  * Erythrocyte sedimentation rate (ESR)
  * Patient assessment of disease activity (VAS; mm)
  The DAS-28 is evaluated using a scale:
  0 - 3.2: low disease activity 3.2 - 5.1: moderate disease activity > 5.1: severe disease activity
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Standard Dose | High Dose
Number analyzed (Participants) | 10 | 9
Units on a Scale | 2.87 (0.93) | 2.66 (0.11)

2. Secondary Outcome: HAQ (Health Assessment Questionnaire)
Time Frame: 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Standard Dose | High Dose
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 5/10 | 4/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose (N=10) | High Dose (N=9)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4) — Nausea after the intake of methotrexate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less